CLINICAL TRIAL: NCT04936516
Title: Effectiveness Comparison Between McGrath and C-MAC Video Laryngoscope in Endotracheal Tube Insertion
Brief Title: McGrath vs. C-MAC Video Laryngoscopy Comparison in Endotracheal Tube Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Christopher Ryalino, MD, Principal Investigator, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UNUD-CTR-FK110621-001
Record Dates: First submitted 2021-06-10; First posted 2021-06-23 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Intubation; Difficult or Failed
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McGrath Video Laryngoscope (Active Comparator)
  Interventions: Device: Endotracheal intubation
- C-MAC Video Laryngoscope (Active Comparator)
  Interventions: Device: Endotracheal intubation

INTERVENTIONS:
Device: Endotracheal intubation — Endotracheal intubation using either McGrath or C-MAC video laryngoscopy

SUMMARY:
Tracheal intubation is commonly performed using a standard Macintosh blade, but recently there has been advanced technology using video laryngoscopy (VL).In this modern era, there are various types of available VL to make it easier for anesthesiologists to perform intubation, especially in patients with difficult airway anatomy.

Various studies showed different results regarding the effectiveness of both C-MAC® and McGrath®, by assessing the comparison of the effectiveness, valuable information will be obtained for further consideration by experts in choosing the best tools in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Elective surgery patients without neck and face trauma
2. Undergo surgery requiring general anesthesia with endotracheal intubation
3. Patients with physical status ASA I-III
4. Patients aged 18-65 years
5. Nutritional status (BMI < 35 Kg/m2)

Exclusion Criteria:

1. Patients refusal to be included in the study
2. Patients with cervical spine instability
3. Anatomical and structural abnormalities of the maxillary teeth
4. Thyromental distance <6 cm and inter-incisor distance <3.5 cm
5. History of difficult intubation
6. LEMON criteria ≥ 3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Intubation time | From first intubation attempt until successful intubation, an average of one minute
  Time required to perform intubation until endotracheal tube is properly positioned
Ease of intubation | From first intubation attempt until successful intubation, an average of two minutes
  Difficulty level of intubation, scores 1-2, 1=effortless, 2=difficult

SECONDARY OUTCOMES:
Number of intubation attempts | From first intubation attempt until successful intubation, an average of one minute
  The number of times required for a successful intubation
Glottic visualization | During first intubation attempt, an average of 30 seconds
  Visualization of glottic assessed by the POGO (Percentage of Glottis Opening) score, 1=best, 4=worst
Complications of intubation | From first intubation attempt until successful intubation, an average of one minute
  Includes orotracheal trauma, presence of blood in the blades, laryngospasm, bradycardia

CONTACTS AND LOCATIONS:
Overall Officials: Tjokorda GA Senapathi, Dr, Study Chair — Udayana University; Jhoni P Pasaribu, Study Director — Udayana University; Christopher Ryalino, Principal Investigator — Udayana University
Locations (1):
- Sanglah General Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No